CLINICAL TRIAL: NCT06576336
Title: 3D is Better for Adrenal: a Randomized Clinical Trial About Use of 3D Laparoscopy Versus 2D Laparoscopy in Adrenal Surgery
Brief Title: A Randomized Clinical Trial About Use of 3D Laparoscopy Versus 2D Laparoscopy in Adrenal Surgery
Acronym: 3DAdrenal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Full Professor of Surgery, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D is better
Record Dates: First submitted 2024-08-17; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Adrenal Mass; Adrenal Adenoma; Adrenal Gland Neoplasms
Keywords: adrenal surgery; laparoscopic adrenalectomy
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Adrenal Gland Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D group (Active Comparator): patients underwent to 2D laparoscopic adrenalectomy for adrenal mass.
  Interventions: Procedure: laparoscopic adrenalectomy
- 3D group (Experimental): patients underwent to 3D laparoscopic adrenalectomy for adrenal mass.
  Interventions: Procedure: laparoscopic adrenalectomy

INTERVENTIONS:
Procedure: laparoscopic adrenalectomy — laparoscopic adrenalectomy

SUMMARY:
Comparison between 2D traditional laparoscopic surgery and 3D laparoscopy for adrenal surgery.

DETAILED DESCRIPTION:
Laparoscopic adrenalectomy is today considered the gold standard of treatment for adrenal tumors. This technique was described for the first time by Gagner in 1992 and in the past years several studies have shown the advantages of laparoscopic approach with decrease of the perioperative morbidity, lower complication rates, less operative blood loss, less postoperative pain and shorter hospital stay compared with open adrenalectomy. Laparoscopic surgery is more difficult to learn and requires different psychomotor skills than open laparotomy. In fact, the surgeons have to work in a three-dimensional space, but are guided by two-dimensional images. The development of high definition cameras does not eliminate the major limitation of two-dimensional (2D) laparoscopy: lack of depth perception and lose of spatial orientation with potential increasing the strain for the surgeon, the risk of errors and the operative time. Three-dimensional (3D) HD laparoscopy was developed as an alternative to conventional 2D laparoscopy.

In literature there are still few clinical studies on use of 3D in laparoscopic adrenalectomies with different results.

For these reasons the investigators propose an international multicenter study to compare 3D laparoscopic adrenalectomy with standard laparoscopic adrenalectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients competent to give consent
* aged between 18 and 85 years
* functioning and not functioning benign adrenal lesions,
* adrenal malignancies candidate to laparoscopic adrenal surgery.

Exclusion Criteria:

* open adrenal surgery
* preoperative signs of local periadrenal invasiveness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
periperative surgical outcomes | 30-postoperative days
  evaluation of intraoperative surgical complication during laparoscopic adrenalectomy with YES or NO and questionnaire about resolution of complications. In details the investigators evaluates: vascular complications (Major lesions: renal artery, renal vein; aorta; vena cava; sovrahepatic veins. Minor lesions: adrenal vessels; accessory renal vessels; others); complication hollow viscus (bowel; colonic; stomach; urether); complication parenchymatous viscus (renal; adrenal; spleen; diaphragm); resolution of complications; conversion to open surgery. 30-day postoperative complications (only grade 3 - 4 - 5 sec. Clavien-Dindo classification)

SECONDARY OUTCOMES:
depth perception | intraoperatory time
  evaluation of depth perception during surgical procedure with a questionnaire administered to surgical team with a score from 1 (min depth) to 5 (max depth)
definition of surgical plane | intraoperatory time
  definition of surgical plane during surgery with a questionnaire administered to surgical team with a score from 1 (min definition) to 5 (max definition)
evaluation of surgical strain | intraoperatory time
  variables of surgical strain: wrist, hand, neck, back, dizziness and/or headache (Yes=1; No=0).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Giuseppe Di Buono, Palermo, PA
  - Italy, Palermo

IPD SHARING:
Plan to Share IPD: No
databse is in the possession of the corresponding author and available upon request after publication of research.

REFERENCES:
- [Result] Agrusa A, di Buono G, Chianetta D, Sorce V, Citarrella R, Galia M, Vernuccio L, Romano G, Gulotta G. Three-dimensional (3D) versus two-dimensional (2D) laparoscopic adrenalectomy: A case-control study. Int J Surg. 2016 Apr;28 Suppl 1:S114-7. doi: 10.1016/j.ijsu.2015.12.055. Epub 2015 Dec 18. PMID 26708842